CLINICAL TRIAL: NCT04171583
Title: Characterisation of Mucoid Staphylococcus Aureus Recovered From the Airways of Cystic Fibrosis Patients: Prevalence and Impact on Clinical Course
Brief Title: Mucoid Staphylococcus Aureus in Cystic Fibrosis Airways
Acronym: mucostaph
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Barbara Kahl, Professor, University Hospital Muenster
Other Study IDs: MZM study
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Staphylococcus Aureus Pneumonia; Lung Diseases; Cystic Fibrosis; Lung Function Decreased
Keywords: cystic fibrosis; staphylococcus aureus; mucoid
MeSH Terms: conditions — Pneumonia, Staphylococcal; Lung Diseases; Cystic Fibrosis; Respiratory Insufficiency; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — respiratory specimens: throat swabs, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mucoid S. aureus: CF patients with mucoid S. aureus
- non-mucoid S. aureus: CF patients with non-mucoid S. aureus

SUMMARY:
Recently, the investigators described a new mucoid phenotype of Staphylococcus aureus cultured from the airways of cystic fibrosis (CF) patients.In this observational study, the investigators plan to determine the prevalence of mucoid S. aureus in respiratory specimens of CF patients and a possible impact of mucoid S. aureus on lung disease severity.

DETAILED DESCRIPTION:
S. aureus is one of the first isolated pathogens recovered from the airways of CF patients. In many patients, S. aureus persists for decades in spite of antibiotic treatment and host defence. During persistence in the airways, S. aureus needs to adapt to this hostile niche. Just recently, the investigators described mucoid S. aureus isolates as a so far not reported phenotype recovered from the airways of CF patients. These mucoid isolates carried a 5bp-deletion in a part of the "intercellular adhesion operon (ica) leading to hyper-expression of biofilm. So far, neither the prevalence of mucoid S. aureus nor the impact on lung disease in CF patients is known. The investigators plan to perform a clinical study to determine the prevalence of mucoid S. aureus isolates in a cross-sectional study and the impact of identified mucoid S. aureus on the clinical course of the lung disease by observing patients with mucoid S. aureus for 12 months in comparison with a group of age-, gender- and P. aeruginosa-positive/negative matched group of S. aureus-positive patients without mucoid isolates.

ELIGIBILITY:
Inclusion Criteria:

* CF patients with chronic S. aureus in respiratory specimens (50% positive S. aureus cultures within one or two years before recruitment)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients with chronic S. aureus in respiratory specimens
Sampling Method: Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
lung function of patients with mucoid S. aureus will be compared to age and gender matched patients with only normal S. aureus | one year
  lung function assessed by FEV1% predicted, which is performed during the visits at the cystic fiboris center, will be reported in case report forms to the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Kahl, MD, Principal Investigator — University Hospital Muenster
Locations (13):
- University Hospital Wien, Vienna, Austria
- Germany (12):
  - University Hospital Ruhr University Bochum, Bochum
  - University Hospital Cologne, Cologne
  - Ruhrlandklinik Essen, Essen
  - University Hospital Essen, Essen
  - University Hospital Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - LMU München, München
  - University Hospital Muenster, Münster
  - Clemenshospital, Münster
  - University Hospital Rostock, Rostock
  - University Hospital Tübingen, Tübingen
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rumpf CH, Janssen T, Hait RJ, Romme K, Decker C, Peters J, Czowalla C, Deiwick S, Gorlich D, Dubbers A, Grosse-Onnebrink J, Kessler C, Kuster P, Schultingkemper H, Hebestreit H, Graepler-Mainka U, van Koningsbruggen-Rietschel S, Schildberg T, Renner S, Nahrig S, Wollschlager B, Schlegtendal A, Sutharsan S, Stehling F, Junge S, Ballmann M, Schwartbeck B, Kahl BC. Mucoid Staphylococcus aureus: A Clinical Trial of Its Prevalence and Association with Lung Function in People with Cystic Fibrosis. Am J Respir Crit Care Med. 2025 May;211(5):854-865. doi: 10.1164/rccm.202407-1474OC. PMID 39918841